CLINICAL TRIAL: NCT00412789
Title: A Phase IA, Open-label, Dose Escalation Study of Patupilone Administered Intravenously Every 3 Weeks in Adult Patients With Advanced Solid Tumors
Brief Title: Efficacy and Safety of Patupilone in Patients With Advanced Solid Tumors in Japan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEPO906A1103
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Last update posted 2010-05-31 (Estimated); Status verified 2010-05

CONDITIONS: Tumors
Keywords: Advanced solid tumor; Patupilone
MeSH Terms: conditions — Neoplasms | interventions — epothilone B

ARMS (1):
- EPO906 (Experimental)
  Interventions: Drug: Patupilone

INTERVENTIONS:
Drug: Patupilone
  Other Names: EPO906

SUMMARY:
The study will evaluate the safety and efficacy of Patupilone in adult patients with advanced solid tumors.

ELIGIBILITY:
Inclusion criteria:

* Patients with a histologically/cytologically confirmed diagnosis of advanced solid tumors refractory to or unsuitable for standard therapy, or for whom no standard therapy exists
* Patients with WHO Performance Status of 0-1 ( Karnofsky Performance Status of 80-100)
* At least one measurable lesion

Exclusion criteria:

* Patients with any peripheral neuropathy
* Patients with unresolved diarrhea
* Patients with severe and/or uncontrolled medical conditions or infections that require systemic therapy

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-08; Primary Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Dose-limiting Toxicity | 18 months

SECONDARY OUTCOMES:
Safety and tolerability of patupilone assessed by CTCAE | 18 months
Pharmacokinetic profile of patupilone | 18 months
Anti-tumor activity of patupilone according to the RECIST guidelines | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Tokyo, Japan